CLINICAL TRIAL: NCT01957722
Title: A Phase 3, Prospective, Randomized, Partially Blinded Multi-Center Study to Measure the Safety and Efficacy of NOVOCART 3D Compared ot Microfracture in the Treatment of Articular Cartilage Defects
Brief Title: NOVOCART®3D for Treatment of Articular Cartilage of the Knee
Acronym: N3D
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aesculap Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-1220
Record Dates: First submitted 2013-09-17; First posted 2013-10-08 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Articular Cartilage of the Femoral Condyle Between 2-6cm2
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NOVOCART 3D (Experimental): Scaffold assisted autologous chondrocyte Implant
  Interventions: Biological: NOVOCART 3D
- Microfracture (Active Comparator): considered a typical treatment for articular cartilage repair
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: Microfracture — Surgical procedure which creates a marrow clot in the prepare cartilage defect.
  Arms: Microfracture
Biological: NOVOCART 3D — combination product- biologic (autologous chondrocytes) /device (scaffold) implant
  Arms: NOVOCART 3D

SUMMARY:
This study is to compare NOVOCART 3D relative to Microfracture for the treatment of knee cartilage defects. Efficacy will be evaluated by both pain and function. Safety will also be evaluated.

DETAILED DESCRIPTION:
Subjects with articular knee defects will be randomized to receive either Microfracture or NOVOCART 3D. Subjects will be followed for five years in total and will be evaluated for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Isolated articular cartilage lesions on the femoral condyle 2-6 cm2
* Minimum score on the KOOS questionnaire

Exclusion Criteria:

* Instability of the knee joint
* Arthritis
* Autoimmune disease
* Immune suppression
* Prior surgical treatment using mosaicplasty, autologous chondrocyte implantation and/or microfracture (debridement and lavage are acceptable beyond three months from baseline)
* Bone disease
* Any degenerative muscular, connective tissue or neurological condition or other disease process that would interfere with healing or the evaluation of outcome measures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - Pain Subdomain | 24 months post treatment
  As measured by a change in KOOS (pain subdomain) score at 24 months from baseline
Knee injury and Osteoarthritis Outcome Score (KOOS) - Function Subdomain | 24 months post treatment
  As measured by a change in KOOS score (activity of daily living subdomain) at 24 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiro, PhD, Study Director — Octane Biotherapeutics, Inc.
Locations (35):
- United States (30):
  - Grossmont Orthopaedic Medical Group, La Mesa, California
  - UCLA, Los Angeles, California
  - Stanford Medicine, Redwood City, California
  - Cu Sports Medicine, Denver, Colorado
  - Yampa Valley Medical Center, Steamboat Springs, Colorado
  - Tenet Florida Physician Services, Boca Raton, Florida
  - Paley Orthopedic and Spine Institute, West Palm Beach, Florida
  - Saint Alphonsus Medical Group, Meridian, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Tria Orthopaedic Center, Bloomington, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri Healthcare, Columbia, Missouri
  - Mount Sinai Faculty Practice Associates, New York, New York
  - Plancher Orthopaedics & Sports Medicine, New York, New York
  - Long Island Bone and Joint Llp, Port Jefferson, New York
  - Ohio State University Sports Medicine, Columbus, Ohio
  - Tulsa Bone and Joint Associates, Tulsa, Oklahoma
  - St. Luke'S University Health Network, Bethlehem, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny - Singer Research Institute, Pittsburgh, Pennsylvania
  - Clinical Research Solutions, Jackson, Tennessee
  - Alpine Orthopaedics, North Logan, Utah
  - University of Virginia, Charlottesville, Virginia
  - The Orthopaedic Center of Central Virginia Inc, Lynchburg, Virginia
  - Advanced Orthopaedics, Richmond, Virginia
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Simon Fraser Orthopaedic Fund, Surrey, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - St. Josephs Healthcare Hamilton, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario

IPD SHARING:
Plan to Share IPD: No